CLINICAL TRIAL: NCT02409641
Title: A Pilot Study Investigating the Impact of Different IOL Designs on Subjective 2D and 3D Image Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-011214
Record Dates: First submitted 2015-02-24; First posted 2015-04-07 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Lenses; Intraocular Sensitivity; Visual Acuity
Keywords: IOL

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 30 healthy male and female subjects (Experimental): 30 healthy male and female subjects , age 18-35 years
  Interventions: Drug: Cyclopentolatehydrochloride 0,5% eye drops

INTERVENTIONS:
Drug: Cyclopentolatehydrochloride 0,5% eye drops — 1 drop in study eye

SUMMARY:
The WHO, states that age related cataracts account for 51 percent of worldwide blindness and affect about 20 million people. Surgery with intraocular lens (IOL) implantation is the first line treatment for cataracts, thus there is an on going effort to improve IOL design and performance.

It is planned to compare three different IOL designs in a psychophysical test setting. Most IOL testing is done in 2D scenarios such as Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity or contrast sensitivity testing. The use of 3D scenario would allow testing a more real-life situation.

As various downsides of different IOL designs have been reported, testing of IOLs before surgical implantation is a promising approach to maximise patient satisfaction. Known deficiencies include amongst others reduced contrast sensitivity or light intensity.

To test three different IOL designs, it is planned to have 2D healthy young subjects look through a stable, table mounted spectacle frame, in which the different IOLs can be inserted. This allows for subjective testing of IOL's in a 2D and 3D scenario.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings
* Refractive spherical error between between -1 and +1 diopters, refractive cylindrical error between -0,25 and +0,25 diopters
* Dominant eye : right eye ( used as study eye)

Exclusion Criteria:

* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Visual Acuity measured by Early Treatment of Diabetic Retinopathy Study Chart | 1 study day

SECONDARY OUTCOMES:
Contrast Sensitivity measured by Pelli-Robson Contrast Sensitivity Chart | 1 study day

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Schmidl, MD, PhD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria